CLINICAL TRIAL: NCT06260384
Title: Clinical Profile and Current Strategies in Management of Wolf-Parkinson-White Syndrome and Asymptomatic Pre-excitation in Africa (a Multicenter WPW African Registry)
Brief Title: Wolf-Parkinson-White Syndrome and Asymptomatic Pre-excitation in Africa (a Multicenter WPW African Registry)
Status: Recruiting | Type: Observational
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Other Study IDs: FMASU R 139/2022
Record Dates: First submitted 2024-02-07; First posted 2024-02-15 (Actual); Last update posted 2024-02-26 (Actual); Status verified 2024-02

CONDITIONS: Wolf Parkinson White Syndrome; Arrythmias
Keywords: WPW syndrome; ECG; RF ablation; Africa
MeSH Terms: conditions — Wolff-Parkinson-White Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- All patients attending outpatient cardiology clinics or referred for EP study: Participants will be recruited from outpatient cardiology clinics and inpatient cardiology wards at twenty cardiac centers in 17 countries spread across all African regions. They all belong to the Africa Heart Rhythm Association (AFHRA) network, and participants are included if they have a preexcitation (WPW) pattern on an ECG. A written consent will be obtained, and an ethical clearance from each center will be obtained from their institution. The exclusion criteria were a lack of consent.
  Interventions: Other: electrocardiogram

INTERVENTIONS:
Other: electrocardiogram — it is a non-invasive study to diagnose criteria of Wolf-Parkinson-Wall syndrome and detect any arrhythmias

SUMMARY:
The purpose of this prospective observational study is to characterize the clinical profile of patients with WPW syndrome and patients with asymptomatic WPW pattern on ECG in different African countries and how these patients are managed across Africa Participants would include many different ethnicities at centers where the number of cardiac patients treated is high. All patients attending outpatient cardiology clinics or referred to Cath Lab for electrophysiological studies who are diagnosed to have a Wolf-Parkinson white pattern on the ECG are either symptomatic or asymptomatic. All patients fulfilling the eligibility criteria will be approached by the research team and asked if they wish to take part in the study.

The exclusion criteria will be any participant who does not consent to the study.

A baseline cardiovascular history (including hypertension, diabetes, heart failure, coronary artery disease, hyperlipidemia, smoking, valve disease, and arrhythmia) will be recorded.

A detailed history will be taken about symptoms, medications and presence of family history of similar cases or sudden cardiac death 12-lead ECG will be recorded to confirm the presence of pre-excitation and determine the localization of the accessory pathway using the modified Aruda algorithm. This will be done by two of the research teams in each center.

Then other data from the electrophysiological study and ablation will be filled in by the research team from the data systems of each center.

DETAILED DESCRIPTION:
A specifically designed electronic report is used and includes the patient's baseline characteristics, symptoms if present, presence of underlying heart disease, family history of any similar conditions, or sudden cardiac death (SCD).

ECG analysis will be done for criteria of WPW pattern, localization of the site of the accessory pathway, and the algorithm used for that; all will be recorded.

Our sample is divided according to clinical presentation into patients with WPW syndrome (those with symptoms or documented tachycardia) and asymptomatic subjects (ventricular pre-excitation on ECG without symptoms).

In patients with WPW syndrome, data will be collected, including symptoms, type of documented tachyarrhythmia, acute management of this arrhythmia on time, and the long-term management strategy, either pharmacological or interventional therapy.

In patients who are referred for electrophysiological (EP) study for mapping and radiofrequency (RF) catheter ablation, all data are recorded, including the method of the study, either fluoroscopic guided or three-dimensional (3D mapping), acute success, site of successful ablation, complications, and long-term success after a one-year follow-up.

Regarding asymptomatic subjects, we collect data on risk stratification, either a noninvasive assessment like a stress electrocardiogram or an invasive electrophysiological (EP) study, and allowance to do exercise and practice sports.

At the end of the study, the performance of each center regarding the management strategy for WPW syndrome was assessed blindly by two European heart rhythm association (EHRA) certified experts in electrophysiology field based on the recent published guidelines of European society of cardiology (ESC).

Socio-economic determinants and health metrics such as the human development index (HDI), health expenditure as a percentage of the gross demographic product (GDP), and the effective health coverage index (UHC) will be compiled together with the EP procedure density of each center to determine the impact of health governance in the management of patients with cardiac pre-excitation. EP procedure density is defined as the ratio between the number of procedures and the years of experience of the index center.

ELIGIBILITY:
Inclusion Criteria:

Patients who have a preexcitation (WPW) pattern on an ECG.

Exclusion Criteria:

any participant who does not consent to the study. Any participants who have structural heart disease History of other arrhythmogenic diseases like Brugada syndrome, Arrhythmogenic AR dysplasia, long QT syndrome..etc Any implantable cardiac rhythm devices

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants are recruited from outpatient cardiology clinics and inpatient cardiology wards at twenty cardiac centers in 17 countries spread across all African regions. They all belong to the Africa Heart Rhythm Association (AFHRA) network, and participants were included if they have preexcitation (WPW) pattern on an ECG either they have symptoms, documented tachyarrhythmias or asymptomatic and accidently discovered
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2022-05-01 (Actual); Primary Completion 2024-05-31 (Estimated); Study Completion 2024-10-31 (Estimated)

PRIMARY OUTCOMES:
No recurrence of symptoms | 12 months
  Disappearance of symptoms after proper management either pharmacological or intervention method based on ESC guidelines on management of supraventricular tachycardia
Assessment of performance outcome of each center | 12 months
  Assessment of quality of management of each shared center in managing the study population based on the recent guidelines

CONTACTS AND LOCATIONS:
Overall Officials: lamyaa E Allam, MD, Principal Investigator — Ain shams university,Cairo
Locations (1):
- Ain shams university, Cairo, Outside US, Egypt

IPD SHARING:
Plan to Share IPD: No
Data will not be shared except the protocol and informed consent at the beginning of the study to keep it safe as researchers are from different countries.
  they all signed an agreement letter for that

REFERENCES:
- [Result] Svendsen JH, Dagres N, Dobreanu D, Bongiorni MG, Marinskis G, Blomstrom-Lundqvist C; Scientific Initiatives Committee, European Heart Rhythm Association. Current strategy for treatment of patients with Wolff-Parkinson-White syndrome and asymptomatic preexcitation in Europe: European Heart Rhythm Association survey. Europace. 2013 May;15(5):750-3. doi: 10.1093/europace/eut094. PMID 23625944
- [Result] Brugada J, Katritsis DG, Arbelo E, Arribas F, Bax JJ, Blomstrom-Lundqvist C, Calkins H, Corrado D, Deftereos SG, Diller GP, Gomez-Doblas JJ, Gorenek B, Grace A, Ho SY, Kaski JC, Kuck KH, Lambiase PD, Sacher F, Sarquella-Brugada G, Suwalski P, Zaza A; ESC Scientific Document Group. 2019 ESC Guidelines for the management of patients with supraventricular tachycardiaThe Task Force for the management of patients with supraventricular tachycardia of the European Society of Cardiology (ESC). Eur Heart J. 2020 Feb 1;41(5):655-720. doi: 10.1093/eurheartj/ehz467. No abstract available. PMID 31504425